CLINICAL TRIAL: NCT06788106
Title: Effect of Different Aerobic Exercise Intensities With Synchronous Music on Psychophysiological, Attentional, Executive Functions and Brain Functional Connectivity Among Medical Students in Jiangsu Province, China
Brief Title: Effect of Aerobic Exercise With Synchronous Music on Functions Among Medical Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Li Le, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/24040378
Record Dates: First submitted 2025-01-02; First posted 2025-01-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Psychological Stress; Aerobic Exercise; Medical Students
Keywords: medical students; mental health; psychophysiological function; attentional function; executive funcion; brain functional connectivity
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): without intervention
- low-intensity with synchronous music group (Experimental): intervened under low-intensity aerobic training with synchronous music of different intensities for 8 weeks, 3 times one week, 40minites one time.
  Interventions: Behavioral: low-intensity aerobic exercise + synchronous music
- medium-intensity with synchronous music group (Experimental): intervened under medium-intensity aerobic training with synchronous music of different intensities for 8 weeks, 3 times one week, 40minites one time.
  Interventions: Behavioral: medium-intensity aerobic exercise + synchronous music
- high-intensity with synchronous music group (Experimental): intervened under high-intensity aerobic training with synchronous music of different intensities for 8 weeks, 3 times one week, 40minites one time.
  Interventions: Behavioral: high-intensity aerobic exercise + synchronous music

INTERVENTIONS:
Behavioral: high-intensity aerobic exercise + synchronous music — This group will be intervened under high-intensity aerobic training with synchronous music for 8 weeks, 3 times every week, 40 minites each time.
  Arms: high-intensity with synchronous music group
Behavioral: medium-intensity aerobic exercise + synchronous music — This group will be intervened under medium-intensity aerobic training with synchronous music for 8 weeks, 3 times every week, 40 minites each time.
  Arms: medium-intensity with synchronous music group
Behavioral: low-intensity aerobic exercise + synchronous music — This group will be intervened under low-intensity aerobic training with synchronous music for 8 weeks, 3 times every week, 40 minites each time.
  Arms: low-intensity with synchronous music group

SUMMARY:
Researchers invite participants to volunteer to participate in this cross-sectional, interventional study. This research examines the effects of 8-week aerobic exercise of different intensities combining synchronized music on psychology, attention, and executive function among Chinese college students, and also validates the reliability and validity of the Chinese version of Brief College Student Hassles Scale, the Perceived Stress Scale for Medical Students, Brief Multidimensional Students'Life Satisfaction Scale, Positive Thinking Skills Scale, Attentional Function Index, Procrastination Assessment Scale-Student and Behavioral Assessment of the Dysexecutive Syndrome-College version, providing a research basis for aerobic exercise to improve the cognitive function and mental health level of Chinese college students. Participants will be invited to participate in the intervention study, in which participants will be assigned to the intervention group and control group. Participation in this study will last approximately 8 weeks for a total of 24 sessions, 40 minutes each session, and participants will not be forced to participate in this study if they do not wish to. This study will include up to 134 participants who will be assigned to the intervention and control groups in a randomized manner.

DETAILED DESCRIPTION:
The study is divided into three parts. Cross sectional study design will be used for Study 1 and Study 2. Experimental study with randomised controlled trial (RCT) will be used for Study 3.

Study-1: Validity and Reliability test of the questionnaire for Chinese population Four scales were selected: the Brief Multidimensional Students' Life Satisfaction Scale - college version (BMSLSS-C), the Positive Thinking Skills Scale (PTSS), Attentional Function Index (AFI), the Executive Functions scale for University settings (UEF).

By using the Brislin (1982) method, firstly, the translation of the questionnaire from English to Chinese first needs to be finished. The translated version needs to be adapted to Chinese culture before implementation. Specifically, a bilingual person will translate all parts of the above questionnaire from English to Chinese. Another bilingual person will translate the translated questionnaire from Chinese into English. The English versions of the two materials will be compared for equivalence, they will be reviewed and finalized by a panel of five experts with experience in sports science, sports psychology, health psychology, and physical education. Then the questionnaire will be distributed through the web-based questionnaire platform.

In the data processing stage, first, the reliability and validity of the three questionnaires will need to be checked, because only with the reliability and validity of the scales, the data will be of analytical value, and the results of the study can be accurately and reliably obtained. For reliability, the magnitude of Cronbach's alpha coefficient, which reflects the degree of internal consistency of the questionnaire, is commonly used as a measure. A Cronbach's alpha coefficient greater than 0.7, according to the general criteria, means that the scale passes the reliability test, and its internal consistency is satisfactory; when the Cronbach's alpha coefficient is greater than 0.8, it means that the scale has good reliability; when the reliability of the scale is below 0.7, the scale needs to be revised at that time. However, in addition to reliability, the validity of the scale needs to be further tested.

Next, validity will be tested using confirmatory factor analysis (CFA) by using Mplus. The CFA model will be constructed separately according to the different dimensions of each scale, the fit indicators for the overall fit measurement were CMIN/DF, RMR, RMSEA, GFI, AGFI, NFI, TLI, and CFI. In addition, the convergent validity of the scale needs to be analyzed. The main indicator of convergent validity is the average variance extracted (AVE), the larger the AVE, the more common the measures are and the better they reflect the same type of problem.

Next, the stability of the translated version of questionnaires employed the test-retest method. An additional 70 participants will be recruited from the 500 participants to re-do the questionnaires after 7 days. This is to compare the stability of the test-retest for the seven questionnaires.

Study-2: Structural equation modeling and path hypothesis validation To test the hypotheses, the full valid sample data are brought into the software Amos, the path hypothesis is tested using the maximum likelihood estimation (ML) method. When using structural equation modeling for model estimation, the overall fit of the model is a test of the extent to which the theoretically constructed conceptual model matches the survey data. The analysis will be conducted using Amos 23.0.

Study-3: Exploring the possible effects of different intensity aerobic training with synchronous music.

Experimental intervention stage, all the selected subjects are divided into four research conditions. Three groups were intervened under aerobic training with synchronous music of different intensities for 8 weeks, and another group served as a control group without intervention. Three aerobic training intervention groups are divided into low-intensity group, moderate-intensity group, and high-intensity group. Defining aerobic training with different intensities based on different MET values. The relationship between MET value and exercise intensity is as follows, less than 3METs belong to low-intensity training, 3-5.9METs belong to moderate-intensity training, greater than 7 METs belong to high-intensity training. The intensity of aerobic training during groups intervention is adjusted through Treadmill Test.

About synchronous music, It is selected using the music tempo according to the exercise intensity as suggested. The music for fast tempo range is 140-150bpm, moderate tempo is 110-120bpm, and slow tempo is 70-80bpm. This study will select 20 pieces of music according to moderate rhythm. After the selection, the 20 songs will be scored by 10 participants using the affect grid and Brunel Music Rating Scale-3, and the highest three song tracks will be selected. To ensure that the intensity of the aerobic exercise is in line with the tempo of the music, we use a DJ beat regulator to do this. When the music plays, the study design and controls for environmental factors are standardized. It is necessary to determine the mode of delivery, frequency /length of time according to the research content when designing music intervention, which is a primary problem on the music variables can be solved. The mode of delivery of music intervention is choose, and the music will be trimmed according to the exercise programme through headphones by the participant.

Before and after intervention, the psychological function, attention, executive function, and brain functional connectivity status of the subjects were evaluated through questionnaires, smartwatch, and Functional near-infrared spectroscopy (fNIRS) brain imaging technology. Then analyze the possible effects of different intensities of aerobic training on the psychological state, attention, and executive function of college students based on the results, as well as the correlation with brain functional connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Medical students willing to participate in aerobic training
* Population of low questionnaire evaluation results
* Subjects achieved a result of 7met or more on the Treadmill Test using the Bruce protocol
* The medical students with low to moderate physical activity level. They are able to exercise, once or twice per week, but are not in the habit of doing so daily

Exclusion Criteria:

* History of major depressive disorder in the past 6 months
* Have a history of alcohol, drug abuse or use of psychiatric drugs
* Have a history of head trauma, neurological disease or other serious illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Psychological function | up to 30 weeks
  Brief Multidimensional Students'Life Satisfaction Scale - college version (BMSLSS-C)
Attentional function | up to 30 weeks
  Attentional Function Index (AFI)
Executive function | up to 30 weeks
  Executive Functions scale for University settings (UEF)
Brain functional connectivity | up to 30 weeks
  Functional near-infrared spectroscopy (fNIRS). Using fNIRS to observe the brain functional connectivity. The fNIRS device used in this experiment was a portable Nir Smart [two wavelengths: 760 and 850 nm, 16 channels (eight light sources and eight detectors); Danyang Huichuang Medical Equipment Co., Ltd., Danyang, China]. According to the 10-20 international standard lead system, the fNIRS helmet was placed on the head of the participant such that the light poles covered the left and right prefrontal areas of the brain, including eight channels of each of the left and right prefrontal lobes (3 × 4 array of emitter and detection light poles).

SECONDARY OUTCOMES:
Positive Thinking Skills | up to 30 weeks
  The Positive Thinking Skills Scale (PTSS)

CONTACTS AND LOCATIONS:
Overall Officials: Garry KP Kuan, PhD, Study Director — Universiti Sains Malaysia
Locations (1):
- Jiangsu Medical College, Yancheng, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Results to be published

REFERENCES:
- [Result] Belkhir Y, Rekik G, Chtourou H, Souissi N. Does warming up with different music tempos affect physical and psychological responses? The evidence from a chronobiological study. J Sports Med Phys Fitness. 2022 Jan;62(1):149-156. doi: 10.23736/S0022-4707.21.12093-6. Epub 2021 Feb 8. PMID 33555672
- [Result] Karageorghis CI, Bigliassi M, Guerin SMR, Delevoye-Turrell Y. Brain mechanisms that underlie music interventions in the exercise domain. Prog Brain Res. 2018;240:109-125. doi: 10.1016/bs.pbr.2018.09.004. Epub 2018 Oct 24. PMID 30390826